CLINICAL TRIAL: NCT02180477
Title: Preliminary Bioequivalence Study of UHAC 62 XX Tablets Compared With a Capsule Formulation
Brief Title: Preliminary Bioequivalence Study of UHAC 62 XX Tablets Compared With a Capsule Formulation in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.251
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- UHAC 62 XX TF1 tablet (Experimental)
  Interventions: Drug: UHAC 62 XX - TF1 tablet; Drug: UHAC 62 XX - TF2 tablet; Drug: UHAC 62 XX - capsules
- UHAC 62 XX TF2 tablet (Experimental)
  Interventions: Drug: UHAC 62 XX - TF1 tablet; Drug: UHAC 62 XX - TF2 tablet; Drug: UHAC 62 XX - capsules
- UHAC 62 XX capsule (Active Comparator)
  Interventions: Drug: UHAC 62 XX - TF1 tablet; Drug: UHAC 62 XX - TF2 tablet; Drug: UHAC 62 XX - capsules

INTERVENTIONS:
Drug: UHAC 62 XX - TF1 tablet
Drug: UHAC 62 XX - TF2 tablet
Drug: UHAC 62 XX - capsules

SUMMARY:
Study to investigate the relative bioavailability of UHAC 62 XX capsule and two different tablet formulations (TF1 and TF2), and to obtain data for rational design of a subsequent pivotal bioequivalence (BE) study between capsule and tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 20 and <= 35 years
* Weight: BMI >= 18.5 and < 25 (Weight (kg) / Height (m²)
* Subjects who are judged by the investigator to be appropriate as the subjects of the study based on results of screening test
* Subjects who volunteer to participate and are able to fully understand and agree with this study by written informed consent

Exclusion Criteria:

* History of gastrointestinal ulcer or surgery of gastrointestinal tract (except appendectomy)
* History of hypersensitivity to meloxicam and/or salicylate (aspirin) and/or Non-steroidal anti-inflammatory drugs (NSAIDs)
* History of aspirin induced asthma (bronchial asthma induced by NSAIDs)
* History of alcohol or drug abuse
* Participation to another trial with an investigational drug within 4 months prior to the administration
* Whole blood donation more than 400 ml within 3 months prior to the administration
* Whole blood donation more than 100 ml within 1 month prior to the administration
* Donation of constituent of blood of more than 400 ml within 1 month prior to the administration
* Any medication within 10 days prior to the administration
* Excessive physical activities within 7 days prior to the administration
* Alcohol drinking within 3 days prior to the administration
* History of orthostatic hypotension, fainting spells or blackouts
* Other than above, those who are judged by the investigator to be inappropriate as the subjects of the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2001-11; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed concentration in plasma) | up to 72 hours after administration
AUC 0-72hr (Area under the concentration-time curve in plasma from zero time to 72 hours) | up to 72 hours after administration

SECONDARY OUTCOMES:
tmax (Time to reach maximum concentration) | up to 72 hours after administration
t1/2 (Terminal half-life in plasma) | up to 72 hours after administration
AUC 0-infinity (Area under the concentration-time curve in plasma from zero time to infinity) | up to 72 hours after administration
MRT 0-t (Mean residence time in the body from zero time to the time of the last quantifiable drug concentration) | up to 72 hours after administration
Number of patients with adverse events | up to 14 days after last administration